CLINICAL TRIAL: NCT07332572
Title: COMPARISON OF INTRAVENOUS DEXMEDETOMEDINE AND TRAMADOL FOR POST OPERATIVE SHIVERING AFTER SPINAL ANESTHESIA FOR CAESAREAN SECTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liaquat National Hospital & Medical College (Other)
Responsible Party: Principal Investigator, Shavez Noor, Shavez Noor, Liaquat National Hospital & Medical College
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LNH
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Shivering Caused by Spinal Anesthesia
Keywords: Shivering
MeSH Terms: interventions — Tramadol; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tramadol group (Active Comparator): Tramadol
  Interventions: Drug: Tramadol; Drug: Dexmedetomidine
- Dexmedetomidine group (Active Comparator): Dexmedetomedine group
  Interventions: Drug: Tramadol; Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Tramadol — Comparative study of tramadol with dexmedetomedine
Drug: Dexmedetomidine — comparative study of tramadol and dexmed

SUMMARY:
To compare the mean time of cessation of post-operative shivering after receiving intravenous dexmedetomidine versus tramadol in patients undergoing caesarean delivery under spinal anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Grade 3 or 4 Shivering

Exclusion Criteria:

* Hypothyroidism
* Known allergies to drugs

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Females who are pregnant
Enrollment: 100 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
SHIVERING TIME | 6 months
  Will assess the cessation time between two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Liaquat National Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided